CLINICAL TRIAL: NCT00183781
Title: Adapting to HIV Disease - A Family Intervention
Brief Title: Effectiveness of a Telephone Intervention Program in Improving Depression, Coping, and Family Functioning in HIV-Infected Individuals and Caregivers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Michael Stein, M.D./Principal Investigator, RI Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063051 (NIH); R01MH063051 (NIH); DAHBR AZ-A
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections
Keywords: HIV; Telephone intervention
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: FITT: Family Intervention - Telephone Tracking

SUMMARY:
This study will evaluate the effectiveness of the Family Intervention: Telephone Tracking (FITT) program in improving depression, coping, and family functioning in HIV-infected individuals and their caregivers.

DETAILED DESCRIPTION:
Individuals who are newly diagnosed with HIV often experience a variety of social and psychological problems, which can leave them depressed and unable to cope with their disease. The complex financial, legal, and psychiatric issues that many HIV-infected individuals must face can be stressful and can negatively affect their health; they may miss doctors' appointments or fail to adhere to a strict HIV medication regimen. The combination of stress and inconsistent medical care can affect the immune system and potentially worsen HIV symptoms.

Because of the multitude of stressors associated with HIV, HIV-infected individuals often rely on a network of family and friends for support; these caregivers, however, are often overwhelmed by their caregiver roles. They may experience helplessness, fear, and depression as a result of their added responsibilities. Family Intervention: Telephone Tracking (FITT) is a telephone-based intervention program that assists in identifying problems and resolving them through referrals to medical and community organizations that provide HIV-related support and services. It is also an educational resource that provides information on the many medical and psychological aspects of HIV infection. The main goal of FITT is to alleviate stress in both the HIV-infected individual and their support network by providing information and resources to help cope with HIV. The purpose of this study is to evaluate the effectiveness of FITT in improving family functioning, enhancing coping skills, and reducing depression in HIV-infected individuals and their caregivers.

This 12-month study will enroll recently diagnosed HIV-infected individuals and one family member or friend who is identified as their primary caregiver. Each pair will be randomly assigned to either the FITT intervention group or to an assessment-only group that will not receive FITT. Individuals who are assigned to receive FITT will utilize the service for Months 1 through 6. HIV-infected participants in both groups will also receive regular medical care throughout the study. Outcome measurements will include self-assessments of depression, coping, and family functioning. In addition, participants receiving FITT will be asked to evaluate the effectiveness of the telephone intervention. All measurements will be assessed at baseline, and Months 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Recently began HIV care
* Currently undergoing HIV care in one of the BRUNAP clinics
* Ability to co-enroll with a primary HIV informal caregiver
* English- or Spanish-speaking

Exclusion Criteria:

* Schizophrenia
* Lacks regular access to a telephone to receive calls

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2000-09; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Decreased depression; measured at baseline, and Months 3, 6, and 12
Improved coping; measured at baseline, and Months 3, 6, and 12
Improved family functioning; measured at baseline, and Months 3, 6, and 12

SECONDARY OUTCOMES:
Efficacy of FITT intervention; measured at baseline, and Months 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Rhode Island Hospital; Penelope Dennehy, MD, Study Director — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Pirraglia PA, Bishop D, Herman DS, Trisvan E, Lopez RA, Torgersen CS, Van Hof AM, Anderson BJ, Miller I, Stein MD. Caregiver burden and depression among informal caregivers of HIV-infected individuals. J Gen Intern Med. 2005 Jun;20(6):510-4. doi: 10.1111/j.1525-1497.2005.0073.x. PMID 15987325
- [Background] Stein M, Herman DS, Trisvan E, Pirraglia P, Engler P, Anderson BJ. Alcohol use and sexual risk behavior among human immunodeficiency virus-positive persons. Alcohol Clin Exp Res. 2005 May;29(5):837-43. doi: 10.1097/01.alc.0000164363.40533.e0. PMID 15897729